CLINICAL TRIAL: NCT01862419
Title: An Electronic Alert System for In-Hospital Acute Kidney Injury: A Randomized, Controlled Trial
Brief Title: An Electronic Alert System for In-Hospital Acute Kidney Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 817822
Record Dates: First submitted 2013-05-16; First posted 2013-05-24 (Estimated); Results first posted 2015-03-25 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2014-04

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alert (Experimental): Text page sent to patient's covering provider and unit pharmacist informing them of the presence of AKI as detected by changes in serum creatinine.
  Interventions: Other: Alert
- Usual Care (No Intervention): Usual care arm. No alert will be provided to the patient's covering provider or unit pharmacist.

INTERVENTIONS:
Other: Alert
  Other Names: Text page sent to patient's covering provider and unit pharmacist informing them of the presence of AKI as detected by changes in serum creatinine.
  Arms: Alert

SUMMARY:
This study will randomize hospitalized patients with acute kidney injury (AKI) to usual care, or an electronic alert intervention. The electronic alert will be in the form of a text page that will be sent to the covering clinician and unit pharmacist once per patient with AKI at the time lab results are uploaded. The investigators hypothesize that such an alert will improve outcomes in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults >=18 years
* Admitted to the Hospital of the University of Pennsylvania for greater than 24 hours.

Exclusion Criteria:

* Dialysis order within 24 hours of admission
* Dialysis order prior to AKI onset
* Initial creatinine >=4.0mg/dl
* Prior admission in which patient was randomized.
* Nephrectomy during the admission
* Admission to hospice service
* Admission to observation status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2393 (Actual)
Dates: Start 2013-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry Fuchs, MD, Principal Investigator — University of Pennsylvania; Francis P Wilson, MD MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Phiadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Wilson FP, Shashaty M, Testani J, Aqeel I, Borovskiy Y, Ellenberg SS, Feldman HI, Fernandez H, Gitelman Y, Lin J, Negoianu D, Parikh CR, Reese PP, Urbani R, Fuchs B. Automated, electronic alerts for acute kidney injury: a single-blind, parallel-group, randomised controlled trial. Lancet. 2015 May 16;385(9981):1966-74. doi: 10.1016/S0140-6736(15)60266-5. Epub 2015 Feb 26. PMID 25726515
- [Derived] Wilson FP, Reese PP, Shashaty MG, Ellenberg SS, Gitelman Y, Bansal AD, Urbani R, Feldman HI, Fuchs B. A trial of in-hospital, electronic alerts for acute kidney injury: design and rationale. Clin Trials. 2014 Oct;11(5):521-9. doi: 10.1177/1740774514542619. Epub 2014 Jul 14. PMID 25023200

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alert | Usual Care
Started | 1201 | 1192
Completed | 1201 | 1192
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alert | Usual Care | Total
Number analyzed (Participants) | 1201 | 1192 | 2393
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (17) | 61 (16) | 60 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 531 | 537 | 1068
  Male | 670 | 655 | 1325
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 38 | 71
  Not Hispanic or Latino | 1168 | 1154 | 2322
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 4 | 6
  Asian | 15 | 30 | 45
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 324 | 323 | 647
  White | 689 | 675 | 1364
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 170 | 159 | 329
Baseline Creatinine [Median (Inter-Quartile Range); unit: mg/dl] | 0.91 [0.60 to 1.37] | 0.90 [0.56 to 1.36] | 0.90 [0.59 to 1.37]
Diabetes [Number; unit: participants] | 352 | 370 | 722

OUTCOME MEASURES:

1. Primary Outcome: Dialysis Within 7 Days
Description: This metric will be sequentially ranked. The provision of acute dialysis therapy will be ranked as a more severe outcome than the worst relative change in creatinine and death will be ranked as a more severe outcome than dialysis.
Time Frame: From start of AKI to 7 days later
Measure: Number; unit: participants
Arm/Group | Alert | Usual Care
Number analyzed (Participants) | 1201 | 1192
participants | 87 | 70

2. Primary Outcome: Death
Time Frame: 7 days of randomization
Measure: Number; unit: participants
Arm/Group | Alert | Usual Care
Number analyzed (Participants) | 1201 | 1192
participants | 71 | 61

3. Primary Outcome: Relative Maximum Change in Creatinine
Time Frame: 7 days of randomization
Measure: Median (Inter-Quartile Range); unit: relative percent change
Arm/Group | Alert | Usual Care
Number analyzed (Participants) | 1201 | 1192
relative percent change | 0.0 [0.0 to 18.4] | 0.6 [0.0 to 17.5]

ADVERSE EVENTS:
Arm/Group | Alert | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/1201 | 0/1192
Other Adverse Events (participants affected / at risk) | 0/1201 | 0/1192

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No